CLINICAL TRIAL: NCT06393283
Title: The Impact of Diaphragm Training on Dysphagia in Elderly Nursing Home Residents: A Preliminary Study
Brief Title: The Impact of Diaphragm Training on Dysphagia in Elderly Nursing Home Residents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GejiYanglaoyuan
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): Diaphragm Training will be given twice a day and 30min per time.
  Interventions: Behavioral: Diaphragm Training
- the blank group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Behavioral: Diaphragm Training — Diaphragm training includes both active and passive methods. Passive training involves placing weights on the participant's abdomen to provide resistance during breathing. Active training involves instructing participants to practice diaphragmatic breathing techniques.
  Arms: the intervention group

SUMMARY:
The goal of this clinical trial is to explore the Diaphragm Training on swallowing function in Elderly Nursing Home Residents (≥60 year old) with swallowing disorders. It primarily aims to address: the effects of Diaphragm Training on swallowing function and quality of life in Elderly Nursing Home Residents. All participants are divided into 2 groups. The intervention group is required to undergo a continuous three-week (21 days) Diaphragm Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

DETAILED DESCRIPTION:
Diaphragm training for dysphagia in elderly nursing home residents involves exercises and techniques aimed at strengthening the diaphragm muscle to improve swallowing function. Dysphagia, or difficulty swallowing, is common among older adults and can lead to complications such as malnutrition, dehydration, and aspiration pneumonia. Diaphragm training may include breathing exercises, postural adjustments, and swallowing maneuvers designed to enhance coordination and strength in the muscles involved in the swallowing process. By targeting the diaphragm, which plays a crucial role in breathing and swallowing coordination, this training approach aims to alleviate dysphagia symptoms and improve overall swallowing function in elderly nursing home residents, thus enhancing their quality of life and reducing the risk of associated health complications.

The goal of this clinical trial is to explore the Diaphragm Training on swallowing function in Elderly Nursing Home Residents (≥60 year old) with swallowing disorders. It primarily aims to address: the effects of Diaphragm Training on swallowing function and quality of life in Elderly Nursing Home Residents. All participants are divided into 2 groups. The intervention group is required to undergo a continuous three-week (21 days) Diaphragm Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old.
* No hospitalization within the past six months.
* With clear consciousness and able to cooperate with questionnaires and training.
* The elderly people who voluntarily participate and agree to adhere until the end of the study.
* early dysphagia caused by sarcopenia.

Exclusion Criteria:

* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Physical disability.
* Difficulty in mobility.
* Simultaneously receiving other therapies that might influence this study.
* Individuals with a gastrostomy.
* Abnormalities of the oral, pharyngeal, or esophageal structures.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Gugging Swallowing Screen | day 1 and day 21
  The Gugging Swallowing Screen is used to assess dysphagia. The Screen consists of 10 items covering various aspects of swallowing, including oral and pharyngeal muscle function, oral sensation, tongue coordination, and more. The total scores range from 1 to 20, with lower scores indicating more severe dysphagia.

SECONDARY OUTCOMES:
Time consumed in eating | day 1 and day 21
  We require participants to eat a lunch according to their daily intake and habits, and count the time consumed
Swallowing-Related Quality of Life Questionnaire | day 1 and day 21
  The Swallowing-Related Quality of Life Questionnaire (SWAL-QOL) is a validated tool used to assess the impact of swallowing difficulties on quality of life. It is a 44-item questionnaire designed to measure the physical, emotional, and social domains of swallowing-related quality of life.The higher final scores indicate the better life quality. The total score will be converted into a standard percentage
Dysphagia Handicap Index | day 1 and day 21
  Dysphagia Handicap Index is a self-reported questionnaire used to assess the impact of dysphagia on an individual's quality of life. It typically consists of multiple questions related to the physical, functional, and emotional aspects of swallowing difficulties. The total score range varies between 0 and 100. A higher score indicates a greater perceived impact of dysphagia on the individual's quality of life.
Eating Assessment Tool-10 | day 1 and day 21
  Subjective perception of swallowing function was assessed using the Eating Assessment Tool-10 (EAT-10). The EAT-10 comprises 10 questions that assess various aspects of swallowing function. Each question is scored on a scale from 0 to 4, indicating the severity of swallowing difficulty, with 0 for no difficulty and 4 for severe difficulty. Participants could rate it based on the subjective perception. The total score on the EAT-10 ranges from 0 to 40, with higher scores indicating more severe swallowing disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Wi, Study Chair — Site Coordinator of United Medical Group